CLINICAL TRIAL: NCT03011307
Title: Efficacy of Intrathecal Oxytocin to Speed Recovery After Hip Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cessation of funding period prior to completion, due to slow recruitment during the pandemic.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00036246
Record Dates: First submitted 2016-12-16; First posted 2017-01-05 (Estimated); Results first posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin 100 micrograms administered intrathecally
  Interventions: Drug: Oxytocin
- Placebos (Placebo Comparator): Placebo injection administered intrathecally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — spinal injection of oxytocin
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Placebo — spinal injection of placebo
  Other Names: Saline
  Arms: Placebos

SUMMARY:
The purpose of this study is to determine the effect of intrathecal oxytocin on speed of reduction in pain for the first 60 days after hip surgery.

DETAILED DESCRIPTION:
This is a single-center, NIH funded clinical study at Wake Forest Baptist Medical Center. The investigators anticipate that intrathecal oxytocin will speed recovery from pain after major surgery (hip arthroplasty). For this study, the investigators will use a randomized, controlled and blinded study of intrathecal oxytocin in patients scheduled for hip arthroplasty, with primary outcome being the slope of change in pain over the first 60 days following surgery, using growth curve modeling and a ln(time) function.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral, primary total hip replacement
* American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* Pregnancy
* Currently Workman's Comp litigation related to hip replacement
* Taking greater than 100 milligrams of morphine (or equivalent)
* Suffering from a psychotic disorder or a recent psychiatric hospitalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from January 12, 2017 to August 3, 2020 at the Orthopeadic Clinics of Atrium Wake Forest Baptist and Davie County facilities.
Pre-assignment Details: Enrollment occurred greater or equal to 2 weeks prior to surgery. A total of 28 individuals were excluded prior to assignment to groups during the period prior to surgery because of withdrawal of consent (n=25) or cancellation of the planned surgery (n=3).
Groups:
- Placebo: Placebo injection administered intrathecally
  Placebos: spinal injection of placebo
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 50 | 48
Completed | 44 | 46
Not Completed | 6 | 2
Not completed — Did not receive study drug: blood pressure or heart rate instability before spinal injection | 3 | 2
Not completed — Did not receive study drug: unable to place spinal needle | 2 | 0
Not completed — Did not receive study drug: unable to obtain study drug from formulating pharmacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 32 | 56
  >=65 years | 20 | 14 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.7) | 59 (10) | 61 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 46 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 40 | 43 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 46 | 90
Worst daily pain [Mean (Standard Deviation); unit: units on a scale] — From daily diaries completed for 2 weeks prior to surgery in which the participant rated each day the worst pain in the past 24 hours with 0=no pain and 10=worst pain imaginable
  units on a scale | 5.0 (2.9) | 5.8 (2.3) | 5.4 (2.7)
Daily steps [Mean (Standard Deviation); unit: Steps per day] — Steps each day for 2 weeks prior to surgery as measured with an activity monitor
  Steps per day | 6440 (4120) | 6918 (4613) | 6672 (4511)
Disability [Mean (Standard Deviation); unit: units on a scale] — Preoperative measure of disability on the World Health Organization Disability Assessment Scale 2.0 where no disability = 12 and severe disability =36
  units on a scale | 20.8 (6.1) | 21.6 (5.0) | 21.2 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Adjusted Trajectory Model for Pain Between Oxytocin and Placebo--Intercept
Description: Daily pain intensity report for each subject was fitted using growth curve model with parameters of intercept (modeled initial pain) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately. The daily pain intensity was the WORST pain (not the average pain) in the past 24 hr on a scale where 0 is no pain and 10 is worst imaginable pain.
  Values represent an intercept of modeled worst daily pain on the first day after hospital discharge across all participants, extracted from the mixed effect model. The intercept is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: The first day after hospital discharge
Measure: Number (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
score on a scale | 8.5 [5.8 to 11.2] | 8.6 [5.9 to 11.3]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; The estimates were conducted using a linear mixed effects model contrasting differences in the oxytocin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline pain, baseline opioid use, age, sex, baseline PROMIS depression and number of other painful conditions; Test type: Superiority — A likelihood-ratio test for change in pain was conducted for each outcome comparing a model with and without oxytocin treatment group. A statistically significant result is interpreted as evidence to support that the oxytocin treatment impacts some element of change after surgery (i.e, intercept or slope); p = 0.75, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Intercept Difference in score on a scale = 0.1, 95% CI 2-sided [0 to .2]

2. Primary Outcome: Comparison of Adjusted Trajectory Model for Pain Between Oxytocin and Placebo--Slope
Description: Daily pain intensity report for each subject was fitted using growth curve model with parameters of intercept (modeled initial pain) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately. The daily pain intensity was the WORST pain in the past 24 hr on a scale where 0 is no pain and 10 is worst imaginable pain.
  Slope is defined as change in pain . Values represent the slope of modeled worst daily pain (0-10 scale as described above) divided by the natural log of time (days) across all participants, extracted from the mixed effect model. The slope is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: Postoperative Day 1 through Postoperative Day 60
Measure: Number (95% Confidence Interval); unit: Score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
Score on a scale | -1.9 [-2.2 to -1.6] | -2 [-2.3 to -1.7]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.057, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Slope Difference = 0.1, 95% CI 2-sided [0.0 to 0.2]

3. Secondary Outcome: Comparison of Adjusted Trajectory Model for Daily Steps Between Oxytocin and Placebo--Intercept
Description: Daily steps for each subject were fitted using growth curve model with parameters of intercept (modeled initial steps) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately. This is considered as the modeled change in activity listed in the protocol.
  Values represent an intercept of modeled daily steps on the first day after hospital discharge across all participants, extracted from the mixed effect model. The intercept is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: The first day after hospital discharge
Measure: Number (95% Confidence Interval); unit: Daily Steps
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
Daily Steps | 144 [-2436 to 3527] | 546 [-3241 to 4332]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.41, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Intercept Difference in Daily Steps = -402, 95% CI 2-sided [-1358 to 553]

4. Secondary Outcome: Comparison of Adjusted Trajectory Model for Daily Steps Between Oxytocin and Placebo--Slope
Description: Daily steps for each subject were fitted using growth curve model with parameters of intercept (modeled initial steps) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately. This is considered as the modeled change in activity listed in the protocol. Values represent the slope of daily steps divided by the natural log of time (days) across all participants, extracted from the mixed effect model. The slope is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: Postoperative Day 1 through Postoperative Day 60
Measure: Number (95% Confidence Interval); unit: Daily steps
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
Daily steps | 562 [-130 to 1248] | 218 [-472 to 907]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; The estimates were conducted using a linear mixed effects model contrasting differences in the oxytocin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline pain, baseline opioid use, age, sex, baseline PROMIS depression and number of other painful conditions. The slope is the number of daily steps divided by the natural log of time in days; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Slope Difference — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Mean Difference (Final Values) = 344, 95% CI 2-sided [173 to 515]

5. Secondary Outcome: Comparison of Adjusted Trajectory Model for World Health Organization Disability Assessment Score 2.0 Value Between Oxytocin and Placebo--Intercept
Description: Weekly World Health Organization Disability Assessment Score 2.0 (WHODAS 2.0) value for each subject was fitted using growth curve model with parameters of intercept (modeled initial score) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately. Scale is 12 to 36 with higher scores meaning greater disability.
  Values represent an intercept of modeled WHODAS 2.0 score one week after hospital discharge across all participants, extracted from the mixed effect model. The intercept is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: Modeled WHODAS 2.0 one week after hospital discharge
Population: The estimates were conducted using a linear mixed effects model contrasting differences in the oxytocin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline World Health Organization Disability Assessment Score 2.0 value, baseline opioid use, age, sex, baseline PROMIS depression and number of other painful conditions.
Measure: Number (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
score on a scale | 23.2 [9.5 to 41.2] | 29.1 [13.5 to 44.8]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; The estimates were conducted using a linear mixed effects model contrasting differences in the oxytocin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline World Health Organization Disability Assessment Score 2.0 value, baseline opioid use, age, sex, baseline PROMIS depression and number of other painful conditions; Test type: Superiority — A likelihood-ratio test for change in World Health Organization Disability Assessment Score 2.0 value was conducted for each outcome comparing a model with and without oxytocin treatment group. A statistically significant result is interpreted as evidence to support that the oxytocin treatment impacts some element of change after surgery (i.e, intercept or slope); p = 0.002, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Intercept Difference: score on a scale = -5.9, 95% CI 2-sided [-9.5 to -2.3]

6. Secondary Outcome: Comparison of Adjusted Trajectory Model for World Health Organization Disability Assessment Score 2.0 Value Between Oxytocin and Placebo--Slope
Description: Weekly World Health Organization Disability Assessment Score 2.0 (WHODAS 2.0) value for each subject was fitted using growth curve model with parameters of intercept (modeled initial score) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately. Scale is 12 to 36 with higher scores meaning greater disability.
  Values represent the slope of WHODAS 2.0 score divided by the natural log of time (days) across all participants, extracted from the mixed effect model. The slope is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model.
Time Frame: Postoperative Day 7 through Postoperative Day 56
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Score on a scale/ln(days)
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
Score on a scale/ln(days) | -7.1 [-11 to -3.2] | -5.6 [-9.5 to -1.7]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Slope Difference = 1.5, 95% CI 2-sided [0.6 to 2.4]

7. Secondary Outcome: Comparison of Adjusted Trajectory Model for Probability of Taking Opioids Daily Between Oxytocin and Placebo--Intercept
Description: Daily probability of taking opioids for each subject was fitted using growth curve model with parameters of intercept (modeled initial pain) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately.
  Values represent an intercept of modeled probability of taking opioid, on a 0-1 probability scale, on the first day after hospital discharge across all participants, extracted from the mixed effect model. The intercept is a number representative of all participants in the Arm and is an estimate with standard deviation based on the model.
Time Frame: The first day after hospital discharge
Measure: Number (95% Confidence Interval); unit: Probability of taking opioids
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
Probability of taking opioids | 0.9995 [0.9985 to 1.0005] | 0.9998 [0.9989 to 1.0007]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; The estimates were conducted using a linear mixed effects model contrasting differences in the oxytocin group versus placebo. In all cases, these differences are adjusted for prognostic variables including baseline opioid use, age, sex, baseline PROMIS depression and number of other painful conditions; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.537, Intercept difference: Opioid probability — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Mean Difference (Final Values) = 0.00035, 95% CI 2-sided [-.00085 to .0015]

8. Secondary Outcome: Comparison of Adjusted Trajectory Model for Probability of Taking Opioids Daily Between Oxytocin and Placebo--Slope
Description: Daily probability of taking opioids for each subject was fitted using growth curve model with parameters of intercept (modeled initial pain) and slope of change in natural log of time, adjusted for prognostic predictors for oxytocin and placebo group separately.
  Values represent the slope of daily probability of taking opioids divided by the natural log of time (days) across all participants, extracted from the mixed effect model. The slope is a number representative of all participants in the Arm and is an estimate with confidence limits based on the model
Time Frame: Postoperative Day 1 through Postoperative Day 60
Measure: Number (95% Confidence Interval); unit: Probability of taking opioids/ln(days)
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
Probability of taking opioids/ln(days) | -0.953 [-0.959 to -0.947] | -0.787 [-0.799 to -0.775]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.010, Mixed Models Analysis — P value not adjusted for multiple comparisons, with threshold of statistical significance set at <0.05; Slope Difference: Opioid probability = -0.166, 95% CI 2-sided [-0.172 to -0.160]

9. Secondary Outcome: Iowa Gambling Task
Description: This is a computer based card game which assesses risk taking and impulsivity in which a score of -100 to 100 is calculated. Lower numbers indicate greater impulsiivity
Time Frame: Preoperative, 2 months after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
units on a scale
  Preoperative | 13 (30) | 21 (31)
  2 Months postoperative | 20 (38) | 22 (37)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Scores were compared statistically at baseline and 2 months between groups using a generalized linear model with time as a fixed factor; Test type: Superiority; p = .55, Regression, Linear; Mean Difference (Net) = 3, Standard Deviation 14

10. Secondary Outcome: Wisconsin Card Sort Task
Description: This is a physical card sorting game which measures attention to shifts in implicit rules as the game progresses. Perseverative errors are the number of sequential errors when rules of the game shift and reflect dysfunction of attention. This score ranges from 0 to 64 with larger numbers reflecting more dysfunction of attention.
Time Frame: Preoperative, 2 months after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
units on a scale
  Preoperative | 6.3 (4.2) | 6.8 (4.9)
  2 Months postoperatively | 8.4 (4.2) | 7.7 (6.7)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Groups were compared over time from baseline to 2 months using a generalized linear model with time as a fixed factor; Test type: Superiority; p = 0.46, Regression, Linear; Mean Difference (Net) = 1.2, Standard Deviation 2.2

11. Secondary Outcome: Tampa Scale of Kinesiophobia
Description: This 17-question scale assesses the degree of fear of pain from joint movement and is commonly used in orthopedic injury or surgery studies. The scale ranges from 17 to 68 with 17 indicating no fear of movement and 68 indicating severe fear.
Time Frame: Preoperative, 2 months after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 44 | 46
units on a scale
  Preoperative | 37 (4.8) | 38 (4.6)
  2 month postoperative | 36 (3.8) | 36 (5.6)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Groups were compared between preoperative and 2 month postoperative sessions using linear regression with time as a fixed factor; Test type: Superiority; p = 0.38, Regression, Linear; Mean Difference (Final Values) = 0.24, Standard Deviation 0.84

ADVERSE EVENTS:
Time Frame: Deaths and Serious adverse events were evaluated from baseline through month 6. Non-serious adverse events were evaluated from baseline through month 2.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/46

LIMITATIONS AND CAVEATS:
The trial was terminated early because of depletion of funding. Power analysis was based on 120 subjects and only 90 were studied before termination of funding .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03011307/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT03011307/SAP_001.pdf
  • Informed Consent Form (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT03011307/ICF_002.pdf